CLINICAL TRIAL: NCT05270096
Title: International Concerted Action to Allocate Children, Adolescents and Young Adults With Relapsed and Refractory Leukemia/Lymphoma to the Right Therapy.
Brief Title: International Leukemia Target Board
Acronym: iLTB
Status: Recruiting | Type: Observational
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: MH21ILT, CRC 2019-062
Record Dates: First submitted 2022-02-15; First posted 2022-03-08 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-10

CONDITIONS: Relapsed Hematologic Malignancy; Refractory Hematologic Malignancy
Keywords: Tumor board; Relapsed leukemia; Treatment prioritization
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia | interventions — Counseling

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Relapsed leukemia: T-ALL:
  First relapse with high MRD after re-induction Newly diagnosed with high MRD after consolidation
  B-ALL:
  1st relapse high risk group, Second or higher relapse, post CAR-T or post HSCT
  AML:
  Second or higher relapse
  Interventions: Other: Advice

INTERVENTIONS:
Other: Advice — non-interventional study

SUMMARY:
The iLTB is a proof-of-concept initiative for children with r/r hematological malignancies, in which available treatment options will be prioritized by actionable events in a harmonized and uniform setting across Europe by a team of biologists, bio-statisticians, bio-informaticians, disease experts, geneticists, flow-experts, clinical trial physicians and also the treating physician.

The iLTB will discuss molecular (genetic lesions), immunophenotypic/surface antigen markers information and, if available, drug response profiles to prioritize these events taking into account the treatment history and treatment intention (bridging to hematopoietic stem cell transplanation/CAR-T or palliative) of each patient followed by a registry to monitor how often iLTB advice has been followed, which other therapy was chosen (off-label, compassionate use) and what the patient outcome is at an aggregated level.

As such the iLTB is non-interventional as it mainly provides advice and registers data on patients discussed in the iLTB.

DETAILED DESCRIPTION:
Improvements in outcome for pediatric hematological malignancies have mainly been driven by the optimization of multi-agent chemotherapy regimens, minimal residual disease monitoring, and risk group stratification based on (cyto)genetic prognostic markers. The prognosis after (multiple) relapse(s) or other new relapsed/refractory (r/r) entities, such as relapse post CAR T-cell therapy in B-cell precursor acute lymphoblastic leukemia (BCP-ALL) and persistent MRD after reinduction therapy for relapsed T-cell ALL, remains poor. This is due to the lack of effective salvage therapies. The options for salvage therapies also differ per disease type: limited options exist in r/r acute myeloid leukemia (AML), T-cell acute lymphoid leukemia and lymphoblastic lymphomas (LBL) compared to r/r BCP-ALL. Recently, new ALL relapse categories have been identified for which an umbrella clinical trial is in development with a molecularly stratified approach: the HEM-iSMART protocol. These new categories consist of multiple relapsed BCP-ALL post CART (which frequently means also post-SCT), and T-ALL/LBL which fail reinduction therapy at first relapse. For AML, early phase clinical studies are set up in the context of the so-called PedAL initiative. Typically second or greater relapsed AML is considered an experimental indication.

Molecular profiling of leukemias and lymphomas is performed in many European countries and the results and potential treatment options are discussed in tumor boards of the national groups. However, numbers in each of these national initiatives are limited, especially when focusing on the new ALL relapse categories, whereas the type of actionable events can be numerous and different between disease types.

The international Leukemia Target Board (iLTB) is fostered by the International Berlin-Frankfurt-Muenster (I-BFM) Resistant Disease and AML committees, the European Inter-group for Childhood Non-Hodgkin Lymphoma (EICNHL) and the ITCC (Innovative Therapies for Children with Cancer in Europe), and has been initiated to discuss these national profiling results with experts from diverse disciplines at a European level, with the aim to better understand the nature of these relapses and to facilitate entry in early phase clinical trials. This will ensure that, as patients are scattered across countries, treating physicians receive the best advice about the prioritization of potential treatment options and open trials according to the patient's actionable events prioritization and treatment history when confronted with these specific relapse situations.

Different from (inter)national tumor boards focused on solid tumors, in addition to the discussion of molecular lesions at the DNA/RNA level, the iLTB will discuss immunophenotypic (CD markers)/surface antigen information and if available centralized drug response profiles (DRP) of r/r hemato-oncology patients for whom standard options for cure are very limited. The available information will be integrated by a newly developed prioritization algorithm that has been developed by an international iLTB development team and which will be optimized prospectively. An actionable event is defined in this study as a tumor characteristic for which targeted therapy is approved, or investigated in a clinical trial for any cancer indication, including but not limited to small molecules and immunotherapy.

It is hypothesized that an international platform for discussing the clinical and biological as-pects of children, adolescents, and young adults with relapsed and refractory hematological malignancies to decide the most appropriate treatment for each individual patient can be a way forward to uniform the community and to tackle these challenges.

The ultimate aim of the iLTB is to improve the outcome of patients with r/r hematological malignancies as defined above by prioritizing actionable lesions in a uniform setting through a panel of experts which advises treating physicians about matching trial(s) or the most appropriate alternative when access to a clinical trial is not possible.

The investigators would like to stress that the iLTB is a platform which is meant to timely share, harmonize, and unify the knowledge about actionable lesions and treatment options for only a subset of r/r cases in Europe, i.e., the patients where the national group asks for discussion in the iLTB, and as such the iLTB does not intend to interfere with outcome evaluations linked to national/local tumor board initiatives.

Enrollment of patients will be coordinated by a representative from the national coordinating center (NCC). Informed consent from the patient to share the data in the iLTB is the responsibility of the treating physician/NCC and is needed prior to discussing the patient's data. Results will be fed back to the treating physician via the NCC or directly.

Treatment interventions however, are not part of this study protocol. Any treatment as a result of iLTB advice will be proposed to the patient by the treating physician and will be subject to a separate consent procedure.

ELIGIBILITY:
Inclusion criteria

1. The patient has been diagnosed with a R/R hematological malignancy;
2. The patient is less than 18 years of age at the time of first diagnosis and less than 25 years at the time of inclusion with relapse/refractory hematological malignancy;
3. The patient is treated in a pediatric/AYA setting or study protocol, with no current standard of care treatment;
4. The patients' life expectancy is at least 6 weeks;
5. The patient has undergone any sort of molecular profiling of his/her tumor and the re-sults of this analysis are available;
6. The patient has undergone flow cytometry in a certified lab and results are available;
7. Written informed consent of patient and/or parent(s)/guardian(s) to discuss the patient in the iLTB according to local law and legislation has been obtained.

Exclusion criteria: none defined

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children less than 18 years of age at the time of first diagnosis and less than 25 years at the time of inclusion with relapsed/refractory ALL, AML or LBL while being treated in a pediatric/AYA center, and for whom no standard of care treatment is available, and for whom molecular and flow cytometry profiling are available for iLTB discussion, and where the national group supports discussing the patient in the iLTB.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-12-31 (Actual); Primary Completion 2030-07-01 (Estimated); Study Completion 2032-06-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients receiving therapy according to the iLTB advice after providing the treating physician with a uniform prioritization of therapy options based on the patient's actionable events. | through study completion, an average of 8 years

SECONDARY OUTCOMES:
Harmonized algorithm to prioritize actionable events options in Europe | through study completion, an average of 8 years
Harmonized algorithm to prioritize treatment options in Europe is available | through study completion, an average of 8 years
Number and frequencies of different types of actionable events reported in the database | through study completion, an average of 8 years
Number of patients being treated with targeted agent according to iLTB advice and compare to previously reported literature by single molecular tumor board initiatives experience | through study completion, an average of 8 years
Calculate the time intervals between time to enrollment, time to recommendation, and time to treatment | through study completion, an average of 8 years
ORR after 1 cycle of treatment of patients with high priority events treated according to the iLTB advice compared to those treated with another therapy (control group) | through study completion, an average of 8 years
Provided reasons by the treating physician why patients were/were not enrolled in trials by 3 monthly follow up | through study completion, an average of 8 years
Assess the OS and EFS of patients discussed in the iLTB | through study completion, an average of 8 years
Analysis and interpretation of the actionable events reported to the iLTB with unmet available clinical trial | through study completion, an average of 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Michel Zwaan, Prof. dr., Principal Investigator — Princess Maxima Center for Pediatric Oncology; Monique den Boer, Prof. dr., Principal Investigator — Princess Maxima Center for Pediatric Oncology
Locations (7):
- UH Gent, Ghent, Belgium
- Righospitalet, Copenhagen, Denmark
- Semmelweis, Budapest, Hungary
- Princess Máxima Center for Pediatric Oncology, Utrecht, Utrecht, Netherlands
- Vall d'Hebron, Barcelona, Spain
- Queen Silvia, Gothenburg, Sweden
- Newcastle Hospital, Newcastle, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All data collected may be shared with third parties by the sponsor following publication of study results, and upon request and a signed material transfer agreement between the third party and the steering committee. Patient privacy and classified information on ongoing trials shall be protected.
Time Frame: After publication
Access Criteria: Request to iLTB steering committee